CLINICAL TRIAL: NCT01508377
Title: Additive Effect of Cognitive Restructuring in a Web-based Treatment for Traumatized Arab People
Brief Title: Effects of an Internet-based Intervention for Posttraumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Berlin Center for the Treatment of Torture Victims (Other)
Responsible Party: Principal Investigator, Christine Knaevelsrud, Clinical Professor, Berlin Center for the Treatment of Torture Victims
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTTV-001
Record Dates: First submitted 2011-12-22; First posted 2012-01-12 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: posttraumatic stress disorder; internet-based psychotherapy; cognitive restructuring; exposure
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cognitive Restructuring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment of PTSD with cognitive restructuring (Experimental): In this arm the PTSD treatment can be divided into three phases.
  First phase: self-confrontation (4 essays)
  Second phase: cognitive restructuring (4 essays)
  Third phase: parting (2 essays)
  Interventions: Behavioral: Exposure for PTSD with cognitive restructuring
- Treatment of PTSD without cognitive restructuring (Experimental): In this arm the PTSD treatment can be divided into only two phases. Compared to the other arm the phase dealing with cognitive restructuring is excluded.
  First phase: self-confrontation (4 essays)
  Second phase: parting (2 essays)
  Interventions: Behavioral: Exposure for PTSD without cognitive restructuring

INTERVENTIONS:
Behavioral: Exposure for PTSD with cognitive restructuring — The treatment lasts five weeks. During that time-frame, participants write ten texts for 45 minutes, twice a week. Each time after having received two texts, the therapists provide feedback and further instructions, which are based upon the manual (Lange et al., 2003)
  The long version of the PTSD treatment (including cognitive restructuring) can be divided into three phases.
  First phase - self-confrontation (4 essays) At the beginning the participants receive psychoeducation about the mechanisms of exposure before writing four essays about their emotionally most painful memories.
  Second phase - cognitive restructuring (4 essays) Again the participants write four texts, however, this time they go beyond mere descriptions and use their experiences to write a supportive letter to an imaginary friend who had been through the same experience.
  Third phase - parting (2 essays) In the third phase, two texts are written in the form of a letter to document the past in a worthy document.
  Arms: Treatment of PTSD with cognitive restructuring
Behavioral: Exposure for PTSD without cognitive restructuring — The treatment lasts five weeks. During that time-frame, participants write ten texts for approximately 45 minutes, twice a week. Each time after having received two texts, the therapists provide feedback and further instructions, which are based upon the manual (Lange et al., 2003).
  The short version of the PTSD treatment can be divided into only two phases. Compared to the long version the phase dealing with cognitive restructuring is excluded.
  First phase - self-confrontation (4 essays) At the beginning the participants receive psychoeducation about the mechanisms of exposure before writing four essays about their emotionally most painful memories.
  Third phase - parting (2 essays) In the third phase, two texts are written in the form of a letter to document the past in a worthy document.
  Arms: Treatment of PTSD without cognitive restructuring

SUMMARY:
For several years now, a very successful treatment of posttraumatic stress disorders has been offered in the Netherlands and in Germany. The contact between clients and therapists takes place exclusively via Internet. The therapists follow a scientifically tested treatment protocol, that defines fixed treatment elements that are adapted to the specific situation of the client. The participants can write at home, in their familiar environment which makes it easier to work on trauma related issues with their therapist. In the last years the treatment was offered in Arabic as well indicating to be an effective treatment for Posttraumatic Stress Disorder (PTSD) in Arabic-speaking countries.

The treatment lasts five weeks. During that time-frame, participants write several texts. The participants decide when they want to write. Each time after having received two texts, the therapists provide feedback and further instructions. The therapists are all trained psychologists, who have received additional training in the interpretation of texts and for the application of the treatment protocol.

The investigators hypothesize that both interventions will significantly improve clinical symptoms of PTSD. Furthermore, the investigators expect improvements in secondary outcomes such as anxiety, depression and quality of life.

DETAILED DESCRIPTION:
Background:

For several years now, a very successful treatment of posttraumatic stress disorders has been offered in the Netherlands and in Germany. The contact between clients and therapists takes place exclusively via Internet. The therapists follow a scientifically tested treatment protocol, that defines fixed treatment elements that are adapted to the specific situation of the client. The participants can write at home, in their familiar environment which makes it easier to work on trauma related issues with their therapist. In the last years the treatment was offered in Arabic as well indicating to be an effective treatment for PTSD in Arabic-speaking countries.

Method:

Traumatized Arabic-speaking participants are allocated at random to a long version (10 sessions) of a manualized writing approach over 6 weeks or to a short version, where the part concerning the cognitive restructuring is excluded. The investigators expect the treatment to be useful for traumatized clients, especially for those who have no access to psychological help otherwise and they hypothesize that both interventions will significantly improve clinical symptoms of PTSD. Furthermore, the investigators expect improvements in secondary outcomes such as anxiety, depression and quality of life. Additionally the investigators are interested, if the short form where the cognitive part is excluded and the focus will be more on confrontation is effective similarly.

Conclusion:

If the interventions prove to be an effective treatment for PTSD in Arabic-speaking countries, the results will lend to support to the establishment of internet-based approaches, especially in countries, where face-to-face therapy cannot be provided. Furthermore a shorter treatment could improve the compliance of the participants, particularly in post-conflict regions where people cannot attend long therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* traumatic experience
* must suffer from posttraumatic stress
* must be fluent in written Arabic
* must have access to the Internet during the treatment

Exclusion Criteria:

* suicidal intentions
* substance abuse
* psychotic experience
* dissociation
* currently receiving psychotherapy elsewhere
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in posttraumatic stress | baseline, post-treatment (1 day after the treatment), 3-months-follow-up (3 months after the treatment)
  Change in Posttraumatic Stress Diagnostic Scale from baseline to post-treatment and 3-months-follow-up

SECONDARY OUTCOMES:
Change in anxiety | baseline, post-treatment (1 day after the treatment), 3-months-follow-up (3 months after the treatment)
  Change in Hopkins Symptom Checklist-25 from baseline to post-treatment and 3-months-follow-up
Change in depression | baseline, post-treatment (1 day after the treatment), 3-months-follow-up (3 months after the treatment)
  Change in Hopkins Symptom Checklist-25 from baseline to post-treatment and 3-months-follow-up
Change in quality of life | baseline, post-treatment (1 day after the treatment), 3-months-follow-up (3 months after the treatment)
  Change in EUROHIS-QOL from baseline to post-treatment and from post-treatment to 3-months-follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Christine Knaevelsrud, PhD, Study Chair — Freie Universität Berlin
Locations (1):
- Treatment Center for Torture Victims Berlin/Freie Universität Berlin, Berlin, Germany

REFERENCES:
- [Derived] Bottche M, Wagner B, Vohringer M, Heinrich M, Stein J, Selmo P, Stammel N, Knaevelsrud C. Is only one cognitive technique also effective? Results from a randomized controlled trial of two different versions of an internet-based cognitive behavioural intervention for post-traumatic stress disorder in Arabic-speaking countries. Eur J Psychotraumatol. 2021 Jul 15;12(1):1943870. doi: 10.1080/20008198.2021.1943870. eCollection 2021. PMID 34345377
- See also: Treatment web-page — http://ilajnafsy.bzfo.de